CLINICAL TRIAL: NCT02586714
Title: Maternal Body Composition Regulates Placental Function
Acronym: MBC
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Nicole Marshall, Primary Investigator, National Center for Research Resources (NCRR)
Other Study IDs: 2KL2RR024141-06 (NIH)
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2015-10

CONDITIONS: Obesity; Pregnancy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal weight
  Interventions: Other: No intervention
- Overweight
  Interventions: Other: No intervention
- Obese
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observation only

SUMMARY:
This study examined the relationships between maternal body composition, placental function, and fetal nutrition and body composition, and sought to determine the most accurate method of maternal body composition analysis in late pregnancy.

DETAILED DESCRIPTION:
This study examined the relationships between maternal body composition, placental function, and fetal nutrition and body composition, and sought to determine the most accurate method of maternal body composition analysis in late pregnancy. This project integrates body composition analysis, nutrition, and metabolic factors to study the impact of maternal body composition and diet on placental function and fetal growth.

Research Project: The proposed enrollment of 41 pregnant women at term (>37 weeks gestation) was completed in September 2013. The subjects underwent four body composition measurements (bioelectrical impedance, skin-fold thickness, BodPod, and deuterium dilution) and dietary surveys along with a fasting blood draw. The subjects returned 2 weeks postpartum for repeat measurements along with a DEXA scan.

ELIGIBILITY:
Inclusion Criteria:

Healthy pregnant women at term with singleton gestation

Exclusion Criteria:

Medical condition requiring daily medication Fetal congenital anomalies Diabetes

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women at term with singleton gestation who were normal weight, overweight, or obese.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Compare maternal body fat measurement | 37 weeks gestation
  Subjects presented for their study visits in the morning following an overnight fast. During the first visit, at 37-38 weeks' gestation, they underwent four measures: 1) ADP, 2) TBW volume by deuterium (2H2O) dilution, 3) skin-fold thickness (SFT), and 4) bioelectrical impedance analysis (BIA). To determine maternal FM (kg) without the presence of the fetus or placenta, and to avoid radiation exposure to the fetus, subjects returned for a second study visit two weeks postpartum for repeat measurements by the above methods plus a dual-energy x-ray absorptiometry scan (DXA) scan. Statistical analysis was performed using the R package Method Comparison Regression, version 1.2.1. Estimates of mean FM (kg) were compared by analysis of variance.

REFERENCES:
- [Derived] Marshall NE, Murphy EJ, King JC, Haas EK, Lim JY, Wiedrick J, Thornburg KL, Purnell JQ. Comparison of multiple methods to measure maternal fat mass in late gestation. Am J Clin Nutr. 2016 Apr;103(4):1055-63. doi: 10.3945/ajcn.115.113464. Epub 2016 Feb 17. PMID 26888714